CLINICAL TRIAL: NCT03327220
Title: A Post-Market, Prospective, Randomized, Controlled Study To Evaluate The Iovera° Device In Treating Pain Associated With Total Knee Arthroplasty
Brief Title: Treatment With Iovera° for Total Knee Arthroplasty (TKA) Post-Operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYO-1265
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: The active group will receive the iovera° treatment prior to a TKA. The control group will receive a TKA and no iovera° treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iovera° Device Treatment Group (Experimental): Iovera° device presurgical cryoneurolysis treatment, 5 (+/- 2) days prior to TKA. Additionally, all participants received treatment as per all the standard pre-, peri-, and post-operative surgical protocols.
  Interventions: Device: iovera°
- Standard of Care Treatment Group (No Intervention): All participants received treatment as per all the standard pre-, peri-, and post-operative surgical protocols.

INTERVENTIONS:
Device: iovera° — The iovera° device applies cold to a target nerve to cause a temporary peripheral nerve block based on a process called Wallerian degeneration (2nd degree axonotmesis) without disrupting connective nerve tissue.
  Arms: iovera° Device Treatment Group

SUMMARY:
This study is designed to investigate whether iovera° treatment prior to TKA decreases cumulative participant opioid use over the course of 6 weeks following TKA while maintaining similar levels of pain relief. The study will also investigate whether there is a relationship between participants treated with iovera° and participant reported pain and function as measured by knee injury and osteoarthritis outcomes score (KOOS JR), numeric rating scale (NRS) for pain; use of hospital services post-TKA and improved physical rehabilitation as measured by range of motion.

ELIGIBILITY:
Inclusion Criteria:

1. 22 to 79 years of age
2. Scheduled to undergo primary unilateral TKA under spinal anesthesia for primary diagnosis of osteoarthritis
3. Participant is a class I-III on the American Society of Anesthesiology (ASA) Physical Classification System
4. Anticipation of discharge to home after inpatient acute post-op phase based on age, co-morbidities, home environment, and social support are in favor of discharge to home in the opinion of the Investigator.
5. Participant is willing and able to give written informed consent.
6. Participant is fluent in verbal and written English.
7. Participant is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
8. Participant is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the participant to an unacceptable risk by study participation.

Exclusion Criteria:

1. Chronic opioid use (defined as daily or almost daily use of opioids for >3 months).
2. Concurrent painful physical condition, surgery, or musculoskeletal disease that requires analgesic treatment during study follow-up that is not strictly related to the target knee being treated with iovera°, which have the potential to confound the postoperative assessments (e.g., significant pain from other joints, chronic neuropathic pain, concurrent or planned contralateral TKA, concurrent foot, neck, spine, hip, or other musculoskeletal disease, arthritis, or planned surgery, etc.).
3. Greater than 15° malalignment (varus or valgus) on pre-operative radiograph.
4. Previous Myoscience treatment.
5. Previous Partial or Total Knee Arthroplasty. Partial or Total Knee Arthroplasty of the contralateral knee is permitted if surgery was completed at least nine (9) months prior to Screening.
6. Body Mass Index ≥ 40
7. Prior surgery in the treatment areas that may alter the anatomy of the infrapatellar branch of the saphenous nerve (ISN) or the anterior femoral cutaneous nerve (AFCN) or result in scar tissue in the treatment area.
8. Any clotting disorder and/or use of an anticoagulant (e.g. warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the device. Low dose aspirin (81mg or less daily) for cardiac prophylaxis allowed.
9. Any local skin condition at the treatment sites that in the Investigator's opinion would adversely affect treatment or outcomes.
10. Open and/or infected wound in the treatment areas.
11. Allergy to lidocaine.
12. History of cryoglobulinemia
13. History of paroxysmal cold hemoglobinuria.
14. History of cold urticaria.
15. History of Raynaud's disease.
16. History of opioid or alcohol abuse.
17. Participant is pregnant or planning to become pregnant while enrolled in the study.
18. Current enrollment in any investigational drug or device study or participation within 30 days prior to screening.
19. Currently being treated for related knee injury under worker's compensation claim or equivalent (i.e. legal case).
20. Any chronic medical condition that in the Investigator's opinion would prevent adequate participation.
21. Any chronic medication use (prescription, over-the-counter, etc.) that in the Investigator's opinion would affect study participation or participant safety.
22. For any reason, in the opinion of the Investigator, the participant may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, etc.).

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Mihalko, MD, PhD, Principal Investigator — UTHSC - COM - Orthopaedic Surgery & Biomedical Engineering
Locations (1):
- Campbell Clinic, Germantown, Tennessee, United States

REFERENCES:
- [Derived] Mihalko WM, Kerkhof AL, Ford MC, Crockarell JR Jr, Harkess JW, Guyton JL. Cryoneurolysis before Total Knee Arthroplasty in Patients With Severe Osteoarthritis for Reduction of Postoperative Pain and Opioid Use in a Single-Center Randomized Controlled Trial. J Arthroplasty. 2021 May;36(5):1590-1598. doi: 10.1016/j.arth.2020.11.013. Epub 2020 Nov 14. PMID 33279353

RESULTS

PARTICIPANT FLOW:
Groups:
- Iovera° Device Treatment Group: Iovera° device presurgical cryoneurolysis treatment, 5 (+/- 2) days prior to total knee arthroplasty (TKA). Additionally, all participants received treatment as per all the standard pre-, peri-, and post-operative surgical protocols.
Period: Overall Study
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
Started | 62 | 62
Safety Population: Received Study Treatment | 59 | 60
Completed | 57 | 58
Not Completed | 5 | 4
Not completed — Adverse Event (AE)/Serious Adverse Event (SAE) | 1 | 2
Not completed — Investigator Decision | 2 | 0
Not completed — Missed Visit 6 (Week 6 Visit) | 0 | 1
Not completed — Fungal infection | 1 | 0
Not completed — Discharged to Rehabilitation | 0 | 1
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.2) | 66.2 (7.1) | 65.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 31 | 26 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 62 | 62 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Participants may have identified as more than one Race.
  participants
    Asian | 1 | 0 | 1
    Black or African American | 10 | 15 | 25
    White | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Opioid Consumption
Description: The cumulative consumption of opioids was determined from the time of Total Knee Arthroplasty (TKA) surgery to 6 weeks post-TKA surgery. Opioid consumption was converted to morphine milligram equivalents (MME) and participant consumption was verified by pill count at follow-up visits. The cumulative morphine equivalent was divided by the number of days to provide the total daily morphine equivalent (TME) for the participant,
Time Frame: From the time of TKA surgery to 6 weeks post-TKA surgery
Population: Intent-to-treat (ITT) population included all participants who were randomized into the study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Error); unit: TME
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
Number analyzed (Participants) | 59 | 60
TME | 4.8 (0.7) | 6.1 (0.7)
Statistical Analysis 1: Comparison: Iovera° Device Treatment Group vs Standard of Care Treatment Group; Testing null hypothesis that true iovera° mean was greater than or equal to the true standard of care mean versus the alternative hypothesis that true iovera° mean was less than true standard of care mean; Test type: Superiority; p = 0.0841, t-test, 1 sided — p-value was calculated from a one-sided, two-sample t-test; Difference in Means = 1.3, 95% CI 2-sided [-0.6 to 3.2]

2. Secondary Outcome: Area Under the Curve (AUC)/Time for Change From Baseline in Knee Injury and Osteoarthritis Outcomes Score (KOOS JR.) Overall Score Through 6 Weeks Post-TKA
Description: The KOOS JR. was a participant completed questionnaire that consists of 7 questions from 3 subscales: stiffness (1 question), pain (4 questions), and function in daily living (2 questions). Standardized answer options are given (5 Likert boxes) and each question was assigned a score from none (0) to extreme (4). A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) was calculated. A positive change from baseline indicates improvement. AUC/time based on Changes from Baseline in KOOS JR. scores through 6 weeks post-TKA, is the AUC of Change in KOOS JR. scores from the Baseline visit through the 6-week visit divided by the number of days from TKA until the 6-week visit. AUC was calculated using the trapezoidal rule and the changes in the KOOS JR. score at the following time points: Baseline (change=0), 72 hours, 2 weeks, and 6 weeks post-TKA.
Time Frame: Baseline to 6 weeks post-TKA surgery
Population: ITT population included all participants who were randomized into the study.
Measure: Mean (Standard Error); unit: score on a scale/days
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
Number analyzed (Participants) | 62 | 62
score on a scale/days | 10.3 (1.6) | 8.4 (1.4)
Statistical Analysis 1: Comparison: Iovera° Device Treatment Group vs Standard of Care Treatment Group; Testing null hypothesis that Standard of Care mean minus the iovera° mean was greater than or equal to non-inferiority margin of 14 versus alternative hypothesis that difference in means was less than 14; Test type: Non-Inferiority — The objective met if the t-test for non-inferiority was statistically significant using a one-sided α = 0.025 level of statistical significance; p < 0.0001, t-test, 1 sided — p-value was calculated from a one-sided, two-sample t-test; Difference in Means = 1.9, 95% CI 2-sided [-2.3 to 6.1]

3. Secondary Outcome: AUC/Time for Change From Baseline in Numeric Rating Scale (NRS) for Pain Through 6 Weeks Post-TKA
Description: NRS was an 11-point scale for self-reporting of pain intensity by participants. Scores range from 0 to 10, where 0 points equals "no pain" and 10 points equals the "worst pain imaginable". A positive change represented improvement (or reduction) in pain intensity. AUC/time based on Changes from Baseline in NRS Pain score through 6 weeks post-TKA, is the AUC of Change in NRS for Pain score from the Baseline visit through the 6-week visit divided by the number of days from TKA until the 6-week visit. AUC was calculated using the trapezoidal rule and the changes in the NRS for Pain score at the following time points: Baseline (change=0), 72 hours, 2 weeks, and 6 weeks post-TKA.
Time Frame: Baseline to 6 weeks post-TKA surgery
Population: ITT population included all participants who were randomized into the study. Overall number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale/days
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
Number analyzed (Participants) | 58 | 59
score on a scale/days
  Pain in The Past 7 Days | 2.2 (2.1) | 1.7 (1.9)
  Pain Right Now | 1.9 (2.7) | 1.5 (2.3)
Statistical Analysis 1: Comparison: Iovera° Device Treatment Group vs Standard of Care Treatment Group; Pain in the Past 7 days - Testing the null hypothesis that the iovera° mean was less than or equal to the Standard of Care mean versus the alternative hypothesis that the iovera° mean was greater than the Standard of Care mean; Test type: Superiority; p = 0.0946, t-test, 1 sided — p-value was calculated from a one-sided, two-sample t-test; Difference in Means = 0.5, 95% CI 2-sided [-0.2 to 1.2]
Statistical Analysis 2: Comparison: Iovera° Device Treatment Group vs Standard of Care Treatment Group; Test type: Superiority — Pain Right Now - Testing the null hypothesis that the iovera° mean was less than or equal to the Standard of Care mean versus the alternative hypothesis that the iovera° mean was greater than the Standard of Care mean; p = 0.2204, t-test, 1 sided — p-value was calculated from a one-sided, two-sample t-test,; Difference in Means = 0.4, 95% CI 2-sided [-0.6 to 1.3]

4. Secondary Outcome: AUC/Time for Change From Baseline in Timed Get Up and Go (TUG) Tests Through 6 Weeks Post-TKA
Description: The time required by the participants to raise from sitting, walk 10 feet, turn around, walk back and sit back down was measured in seconds. A positive change from baseline indicates improvement. AUC/time based on Changes from Baseline in the TUG test through 6 weeks post-TKA, is the AUC of Change in TUG test from the Baseline visit through the 6-week visit divided by the number of days from TKA until the 6-week visit. AUC was calculated using the trapezoidal rule and the changes in the TUG test at the following time points: Baseline (change=0), 72 hours, 2 weeks, and 6 weeks post-TKA.
Time Frame: Baseline to 6 weeks post-TKA surgery
Population: ITT population included all participants who were randomized into the study. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: seconds/days
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
Number analyzed (Participants) | 57 | 59
seconds/days | -1.2 (5.5) | -0.4 (11.3)
Statistical Analysis 1: Comparison: Iovera° Device Treatment Group vs Standard of Care Treatment Group; Testing the null hypothesis that the iovera° mean was less than or equal to the Standard of Care mean versus the alternative hypothesis that the iovera° mean was greater than the Standard of Care mean; Test type: Superiority; p = 0.3231, t-test, 1 sided — p-value was calculated from a one-sided, two-sample t-test; Difference in Means = -0.8, 95% CI 2-sided [-4.0 to 2.5]

ADVERSE EVENTS:
Time Frame: From first treatment up to the end of the study (Up to approximately 12 weeks)
Description: All-cause Mortality: ITT population included all randomized participants. Serious Adverse Events and Adverse Events: Safety population included all participants who received study treatment.
Arm/Group | Iovera° Device Treatment Group | Standard of Care Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 2/59 | 2/60
Other Adverse Events (participants affected / at risk) | 4/59 | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iovera° Device Treatment Group (N=59) | Standard of Care Treatment Group (N=60)
Bilateral Pulmonary Emboli (Vascular disorders) | 1 | 0
R/O Popliteal Arterial Aneurysm (Vascular disorders) | 1 | 0
Neuropsychotic/seizures (Psychiatric disorders) | 1 | 1
Anaphylaxis (Skin and subcutaneous tissue disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iovera° Device Treatment Group (N=59) | Standard of Care Treatment Group (N=60)
R/O Deep vein thrombosis (Vascular disorders) | 4 | 3 — R/O=Rule Out

LIMITATIONS AND CAVEATS:
This study was acquired from another sponsor. Results for the Primary Outcome Measure, Cumulative Opioid Consumption, are reported for the Time Frame (From the time of TKA surgery to 6 weeks post-TKA surgery) because the results for the Time Frame (From the time of hospital discharge to 6 weeks post-TKA surgery) are not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03327220/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03327220/SAP_001.pdf